CLINICAL TRIAL: NCT00940004
Title: TLR Ligand Matured Dendritic Cell Vaccination in Melanoma Patients: the Key Towards a More Potent Immune Induction?
Brief Title: Toll-like Receptor (TLR) Ligand Matured Dendritic Cell Vaccination in Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL22750.000.08; KUN2006-3699
Record Dates: First submitted 2009-06-25; First posted 2009-07-15 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2014-11

CONDITIONS: Melanoma
Keywords: dendritic cell vaccination; melanoma; toll like receptor ligands; vaccines
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cytokine matured DC (Active Comparator): vaccination with autologous dendritic cells matured with standard cytokine cocktail and electroporated with mRNA encoding tumor associated antigens
  Interventions: Biological: autologous dendritic cell vaccination
- TLR ligand matured DC (Experimental): vaccination with autologous TLR-ligand matured dendritic cells electroporated with mRNA encoding tumor associated antigens
  Interventions: Biological: autologous dendritic cell vaccination

INTERVENTIONS:
Biological: autologous dendritic cell vaccination — Autologous monocyte-derived dendritic cells electroporated with mRNA encoding gp100 and tyrosinase and matured with either cytokines or TLR ligands. Dendritic cells are vaccinated intradermal/intravenously 3 times with biweekly intervals every 6 months, if no signs of progression, for a total of 9 vaccinations.

SUMMARY:
Objectives:

This is an exploratory study, consisting of two parts. In part I a dose escalation is performed and the primary objective is the safety of different doses of TLR-dendritic cell (TLR-DC). In part II TLR-DC vaccination will be compared with cytokine-matured DC vaccination and the primary objective of this part is the immunological response to TLR-DC vaccination, with toxicity and clinical efficacy being secondary objectives. These studies will provide important data on the safety and immunological effects of TLR-matured DC.

Study design:

This study is an open label prospective exploratory intervention study.

Study population:

The investigators' study population consists of HLA-A2.1 positive melanoma patients, with proven expression of melanoma associated tumor antigens gp100 and tyrosinase. Melanoma patients with regional lymph node metastasis in whom a radical lymph node dissection is planned or performed within 2 months of inclusion in this study (further referred to as stage III) and melanoma patients with measurable distant metastases (further referred to as stage IV) will be included.

DETAILED DESCRIPTION:
1. Rationale

   Immunotherapy applying ex vivo generated and tumor-antigen-loaded dendritic cells (DC) has now successfully been introduced in the clinic. A limited, but consistent, number of objective immunological and clinical responses have been observed. Thus far it remains unclear why some patients respond and others not, but there is a general consensus that the current protocols applied to generate DC may not result in the induction of optimal Th1 responses. We and others have demonstrated that DC maturation is one of the crucial factors, not only for effective DC migration but also to induce effective anti-tumor immune responses in cancer patients. Currently, the "golden standard" used to mature DC consists of a cocktail of pro-inflammatory cytokines (IL-1beta, IL-6, TNFalpha) and prostaglandin E2 (PGE2). Recent mouse data demonstrated, however, that maturation of DC by solely pro-inflammatory cytokines yielded DC that supported T cell clonal expansion, but failed to efficiently direct effector T cell differentiation. Interestingly, DC matured in the presence of Toll like receptor (TLR) ligands were able to induce full T cell effector function and unleashed more potent immune responses. We recently identified vaccines against infectious diseases that contain TLR ligands and are capable of inducing DC maturation. This knowledge provides a new application for these clinical applicable agents: clinical grade DC stimulators. A clinical grade DC maturation protocol is developed in which TLR ligands (preventive vaccines) and PGE2 are combined which resulted in the generation of mature DC that secrete high levels of the key cytokine IL-12. Moreover, these TLR-ligand matured DC induced T cells secreting at least 20-fold higher levels of the effector cytokines IFNalpha and TNFalpha as compared to DC matured in the absence of TLR ligands. In conclusion, these in vitro data demonstrate that TLR-ligand matured DC are promising candidates to improve immunological and clinical responses in cancer immunotherapy.
2. Objectives

   This is an exploratory study, consisting of two parts. In part I a dose escalation is performed and the primary objective is the safety of different doses of TLR-DC. In part II TLR-DC vaccination will be compared with cytokine-matured DC vaccination and the primary objective of this part is the immunological response to TLR-DC vaccination, with toxicity and clinical efficacy being secondary objectives. These studies will provide important data on the safety and immunological effects of TLR-matured DC.
3. Study design

   This study is an open label prospective exploratory intervention study.
4. Study population

   Our study population consists of HLA-A2.1 positive melanoma patients, with proven expression of melanoma associated tumor antigens gp100 and tyrosinase. Melanoma patients with regional lymph node metastasis in whom a radical lymph node dissection is planned or performed within 2 months of inclusion in this study (further referred to as stage III) and melanoma patients with measurable distant metastases (further referred to as stage IV) will be included.
5. Main study endpoints

The primary objectives of the study are to investigate the toxicity of TLR-DC by dose escalation of DC numbers in part I, and to investigate immunological responses upon TLR-DC vaccination in part II of the study.

Immunological responses are:

1. The migratory capacity of the TLR-ligand matured DC in vivo.
2. The activation of immune cells in vivo.
3. The immunological response induced with TLR-ligand matured DC loaded with mRNA encoding melanoma-associated tumor antigens (gp100 and tyrosinase).

Safety and clinical efficacy are secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* histologically documented evidence of melanoma
* stage III or IV melanoma according to the 2001 AJCC criteria
* HLA-A2.1 phenotype melanoma expressing gp100 (compulsory) and tyrosinase (non- compulsory)
* WHO performance status 0-1 (Karnofsky 100-70)
* life expectancy > 3 months
* age 18-70 years
* no clinical signs or symptoms of CNS metastases
* WBC > 3.0x109/l, lymphocytes > 0.8x109/l, platelets > 100x109/l, serum creatinine < 150 µmol/l, serum bilirubin < 25 µmol/l
* normal serum LDH (< 450 U/l)
* expected adequacy of follow-up
* no pregnant or lactating women
* written informed consent

And in addition for Part I + II:

* stage III melanoma: radical regional lymphnode dissection is planned or performed
* stage IV melanoma: at least one unidimensional measurable target lesions according to RECIST, not previously irradiated, and no significant symptoms of disease requiring other palliative treatments

Exclusion Criteria:

* prior chemotherapy, immunotherapy or radiotherapy < 4 weeks prior to planned vaccination or presence of treatment-related toxicity
* history of any second malignancy in the previous 5 years, with the exception of adequately treated basal cell carcinoma or carcinoma in situ of the cervix serious active infections, HbsAg or HIV positive or autoimmune diseases or organ allografts
* concomitant use of immunosuppressive drugs
* known allergy to shell fish (since it contains KLH)
* rapidly progressive disease
* any serious clinical condition that may interfere with the safe administration of DC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Toxicity of TLR-matured DC (part I) and immunological response upon vaccination with TLR-matured DC (part II) | 3 years

SECONDARY OUTCOMES:
vaccination related toxicity | 5 years
  in terms of local injection site reaction, flu-like symptoms, or otherwise related to vaccination, scored according to CTC version 3.0
clinical efficacy (progression free survival) | 5 years
  time to progression from date of start (apheresis) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: C.J.A. Punt, prof.dr., Principal Investigator — Radboud University Nijmegen Medical Centre, dept of Medical Oncology
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- See also: home page Department of Medical Oncology — http://www.umcn.nl